CLINICAL TRIAL: NCT06641063
Title: Examining the Impact of a Standardized Obstetrics Note Template on Provider Satisfaction, Efficiency, and Perceived Comprehensiveness
Brief Title: Impact of a Standardized Obstetrics Note Template
Status: Recruiting | Type: Observational
Sponsor: MediSys Health Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2223670
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Obstetrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a new standardized obstetrics note template on the quality, efficiency, and provider-perceived comprehensiveness of clinical documentation in a healthcare setting. The investigators aim to determine whether implementing standardized templates improves the completeness, clarity, and accuracy of clinical notes while reducing the time required for healthcare providers to review and document patient encounters.

DETAILED DESCRIPTION:
Clinical documentation is a critical component of patient care, influencing communication among healthcare providers, continuity of care, and overall patient outcomes. Variability in note writing can lead to incomplete or unclear documentation, which may compromise patient safety. Standardized note writing templates have the potential to enhance the quality and efficiency of clinical documentation as well as improve overall provider satisfaction. Research has shown that structured documentation can improve provider efficiency and decrease documentation time. However, little is studied about the implementation of standardized prenatal care visit notes and provider perception of the comprehensiveness of prenatal care and provider satisfaction.

The investigators' study aims to evaluate pre- and post-intervention comparison of questionnaire responses to evaluate changes in the perceived quality and efficiency of clinical documentation. Questionnaires are good for gathering data about abstract ideas or concepts that are otherwise difficult to quantify, such as opinions, attitudes and beliefs. A baseline survey on the current feelings in regards to documentation practices will be collected, followed by the implementation of standardized note writing templates. Post-intervention surveys of the residents will then be gathered to assess the impact of the templates. To ensure an accurate assessment of stakeholders, a response rate of at least 60% (at least 7) is recommended.

This is a pilot longitudinal 4-timepoint panel design monthly survey of Post Graduate Year (PGY)1-4 Obstetrics and Gynecology (OBGYN) residents. The goal of this project is to provide a quality improvement evaluation of the benefits of a new standardized note template for prenatal care visits. Online surveys will be delivered via the Qualtrics survey platform to all residents in the Flushing Hospital Medical Center (FHMC) OBGYN residency program over the course of a 3 month quality improvement initiative. Data will be collected at baseline (immediately prior to the implementation of the note template), 1-month, 2-months, and 3-months.

Primary Outcomes:

* Reduce provider effort in reviewing and documenting prenatal records
* Improve standardization of the documentation and review of prenatal records
* Decrease the time to review patient charts for patient encounters.

Secondary Outcomes:

* Increase confidence in the comprehensiveness of prenatal records
* Increase confidence in the accuracy of prenatal records
* Increase provider satisfaction with the process of reviewing and documenting prenatal records

Procedures:

1. Baseline Data Collection:

   o The baseline survey will be administered to all residents prior to implementation of the standardized note template.
2. Intervention:

   * A training session for all healthcare providers on how to use the standardized templates will be provided during noon conference following baseline survey administration and prior to day one of implementation.
   * The template will be implemented for a predefined period of 3 months, during which the template will be used by all residents for all prenatal encounters.
3. Intervention Evaluation Data Collection:

   o Monthly survey administration will occur during noon-conference during the implementation period at 1-month, 2-months, and 3-months post implementation. The survey will be delivered online via Qualtrics and made accessible to residents during noon-conference via Quick Response (QR) codes and survey links.
4. Data Management and Analysis:

   * After data collection, all survey responses will be immediately de-identified and assigned a unique subject identifier. Subjects will be identified only based on this number and not based on any other personal information or demographic characteristic.
   * To test our primary hypotheses, the investigators will conduct a series of unadjusted and adjusted (i.e., controlling for training year) repeated measures Analysis of Variances (ANOVAs) to evaluate change over time in provider effort, time, confidence, and satisfaction.
   * All analyses will be conducted using Statistical Analysis System (SAS) 9.4 and an alpha level of < .05 will denote statistical significance.

Potential Risks and Benefits:

* Risks: There are minimal risks associated with this study. Participants may experience a learning curve while adapting to the new templates, which could temporarily affect their documentation time.
* Benefits: The study may demonstrate improvements in clinical documentation quality and efficiency, ultimately enhancing patient care and provider satisfaction.

Confidentiality: All data collected will be de-identified to protect participant confidentiality. Data will be stored securely and only accessible to the research team.

Informed Consent: Informed consent will be obtained from all participants prior to their inclusion in the study. Participants will be informed about the study's purpose, procedures, risks, and benefits.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers (physicians, nurse practitioners, physician assistants) at Flushing Hospital Medical Center

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare providers (physicians, nurse practitioners, physician assistants) at Flushing Hospital Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in self-reported effort taken to review and document prenatal notes | From baseline to 3-months

CONTACTS AND LOCATIONS:
Locations (1):
- Flushing Hospital Medical Center, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided